CLINICAL TRIAL: NCT04856969
Title: A Two-arm, Open-label, Single-sequence, Multiple Oral Dosings, Cross-over Design Clinical Trial to Evaluate the Safety and Pharmacokinetic Interaction of ATB-1011 and ATB-1012 in Healthy Adult Volunteers
Brief Title: Clinical Trial to Evaluate Pharmacokinetic Interaction of ATB-1011 and ATB-1012 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autotelicbio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATB-101-001
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — olmesartan; dapagliflozin

STUDY DESIGN:
Intervention Model Description: 2 Intervention group, open, single-sequence, multiple oral administration crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): ATB-1011: 1tab/d for 5days , ATB-1011+ATB-1012: each 1tab/d for 5days
  Interventions: Drug: Olmesartan; Drug: Dapagliflozin
- Arm B (Active Comparator): ATB-1012: 1tab/d for 5days / ATB-1011+ATB-1012: each 1tab/d for 5days
  Interventions: Drug: Olmesartan; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Olmesartan — First stage: ATB-1011 for 5days, repeated administration, Second stage: ATB-1012 + ATB-1011 for 5days, repeated administration
  Other Names: brand name: Olmetec
Drug: Dapagliflozin — First stage: ATB-1012 for 5days, repeated administration, Second stage: ATB-1012 + ATB-1011 for 5days, repeated administration
  Other Names: brand name: Forxiga

SUMMARY:
To evaluate the interaction between two investigational products by comparing and analyzing pharmacokinetic interactions and safety in steady state after multiple oral administration of ATB-1011 or ATB-1012 alone or in combination in healthy adult volunteers.

DETAILED DESCRIPTION:
* Arm A: To evaluate the effect of ATB-1012 on the safety and pharmacokinetic properties of ATB-1011 in steady state.
* Arm B: To evaluate the effect of ATB-1011 on the safety and pharmacokinetic properties of ATB-1012 in steady state.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are over 19 years old at the screening visit
2. Those with a body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 with a weight of 50 kg or more (45 kg or more for women) at the screening visit
3. Those who do not have clinically significant congenital or chronic diseases and have no pathological symptoms or findings upon medical examination at the screening visit
4. Those who determined as suitable study subjects by the principal investigator (or a delegated sub-investigator) in result of planned and conducted laboratory tests such as hematology, blood chemistry, serum, and urine tests according to the characteristics of the investigational product.

Exclusion Criteria:

- 1) Those who have a clinically significant disease or have a history of such disease in the digestive system, cardiovascular system, endocrine system, respiratory system, blood/tumor, infectious diseases, kidney and genitourinary system, mental and nervous system, musculoskeletal system, immune system, otorhinolaryngology, skin system and ophthalmic system.

2) Those who have a history of gastrointestinal surgery (except for simple appendectomy or hernia surgery) that may affect the absorption of drugs or have gastrointestinal diseases 3) Those who have taken drugs that induce and inhibit metabolism enzymes such as barbital drugs within 1 month of the first administration date, or have taken drugs that may interfere with this clinical trial within 10 days of the first administration date. (However, participation is possible depending on the characteristics of pharmacokinetics and pharmacodynamics such as interactions with investigational products or half-life of concomitant drugs) 4) Those who participated in other clinical trials or bioequivalence studies and administered the investigational products within 6 months of the first administration date.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
ATB-1011 AUCτ,ss | 5days, 10days
  the primary endpoints, are converted into natural logarithms, and a point estimate of the difference between the mean values of single and co-administration and 90% confidence intervals thereof is evaluated to evaluate the pharmacokinetic properties.
ATB-1012 AUCτ,ss, | 5days, 10days
  the primary endpoints, are converted into natural logarithms, and a point estimate of the difference between the mean values of single and co-administration and 90% confidence intervals thereof is evaluated to evaluate the pharmacokinetic properties.
ATB-1011 Cmax,ss | 5days, 10days
  the primary endpoints, are converted into natural logarithms, and a point estimate of the difference between the mean values of single and co-administration and 90% confidence intervals thereof is evaluated to evaluate the pharmacokinetic properties.
ATB-1012 Cmax,ss | 5days, 10days
  the primary endpoints, are converted into natural logarithms, and a point estimate of the difference between the mean values of single and co-administration and 90% confidence intervals thereof is evaluated to evaluate the pharmacokinetic properties.

SECONDARY OUTCOMES:
ATB-1011 Tmax,ss | 5days, 10days
  Pharmacokinetic parameters are calculated using a noncompartmental method and descriptive statistics of pharmacokinetic endpoints are presented for each investigational product administration group.
ATB-1011 Cmin,ss | 5days, 10days
  Pharmacokinetic parameters are calculated using a noncompartmental method and descriptive statistics of pharmacokinetic endpoints are presented for each investigational product administration group.
ATB-1012 Tmax,ss | 5days, 10days
  Pharmacokinetic parameters are calculated using a noncompartmental method and descriptive statistics of pharmacokinetic endpoints are presented for each investigational product administration group.
ATB-1012 Cmin,ss | 5days, 10days
  Pharmacokinetic parameters are calculated using a noncompartmental method and descriptive statistics of pharmacokinetic endpoints are presented for each investigational product administration group.

CONTACTS AND LOCATIONS:
Overall Officials: KyungWan Nam, Pharm. D., Principal Investigator — Autotelic.bio
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea